CLINICAL TRIAL: NCT05605717
Title: Non Invasive Evaluation of Liver Fibrosis and Steatosis in Type 2 Diabetic Patient in Assiut University Hospitals
Brief Title: Liver Fibrosis and Steatosis in dm Non Invasive Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed adel mohamed hassan, Resident, Assiut University
Other Study IDs: Liver fibrosis in dm
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre specified group: Fibroscan Abdominal ultrasound Lab investigation
  Interventions: Radiation: Fibroscan

INTERVENTIONS:
Radiation: Fibroscan — Liver fibroscan and ultrasonography
  Other Names: Abdominal ultrasound

SUMMARY:
Non invasive evaluation of liver fibrosis and steatosis in type 2 diabetic patient in Assiut University hospitals

DETAILED DESCRIPTION:
Estimated incidences of non-alcoholic fatty liver disease (NAFLD) all over the world have increased twice in the last two decades, while the incidences of other chronic liver diseases (CLD) have remained unchanged or are on downward trends [LaBrecque ,et al2012]. Traditionally, NAFLD has been reported as a burden condition only in the United States (US) or Western countries. However, nowadays, urbanization has brought about sedentary lifestyles and overnutrition in many Arabian countries, leading to the increase of obesity and metabolic disorders. As the result, NAFLD has been very common . Currently, the population prevalence of NAFLD in the US and Europe is approximately 30 percent{Jian-Gao et al 2017,} Although almost all NAFLD patients have simple steatosis only, 10%20% of patients represent the active form: non-alcoholic steatohepatits (NASH) progressing to liver fibrosis, cirrhosis, heptatocellular carcinoma (HCC) and finally end-stage liver failure [LaBrecque,et al 2012].

NAFLD patients are at 64 times higher risk of cardiovascular disease(CVD), that include coronary artery disease and stroke, than patients without NAFLD [Targher,et al 2016]. Mortality in NAFLD patients is mostly due to CVD events, markedly exceeding the common population{Ekstedt, et al 2006} Type 2 diabetes mellitus (T2DM) is the main risk factor of NAFLD. Patients with T2DM are at a Greater risk of NAFLD and have a higher rate of death and progression to cirrhosis than non-diabetic Individuals [Younossi, et al 2004]. Therefore, screening for NAFLD and evaluating liver fibrosis in the diabetic population is extremely necessary for early detection and management, preventing the progression to advanced fibrosis, cirrhosis and HCC.

NAFLD is diagnosed when there is evidence of ≥ 5% hepatic steatosis either by histology or Imaging and absence of secondary causes of fatty accumulation [Chalasani,et al2018]. FibroScan can assess hepatic steatosis levels, This is a non-invasive, simple-to-perform imaging modality with high accuracy to assess liver stiffness and hepatic fat deposition. Thus far there has been little knowledge on the prevalence of NAFLD and liver fibrosis in diabetic populations in Egypt Therefore our study proposed to estimate the prevalence of NAFLD and the severity of Liver fibrosis by in T2DM patients with the use of fibroscan and other clinical and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with known T2DM or previously unknown diabetes but displaying fasting glucose level of more than 126 mg/dl or HbA1c more than 6.5 % and who were admitted for medical check up, patient divided according to duration of DM to 3 groups less than 5 years from 5 to 10 years and more than 10 years

Exclusion Criteria:

- Patient with Alchole intake,causes of secondary hepatic steatosis abuse of steatogenic drugs(eg: amiodarone,valproic acid ,tetracycline) , positive HBs ag ,HCV ab, measurement failure( marked obesity,ascites,..) or unreliable results on Transient Elastography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samle size was calculated using Epi- Info7, Based on prevelance of NAFLD and type 2 DM all patients In one year the minimum patients required for this study is 60 patient
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis and steatosis in type 2 diabetic patients | 1 year
  our study proposed to estimate the prevalence of NAFLD and the severity of liver fibrosis in T2DM patients taking in account the duration of illness correlation of finding on fibroscan with abnormalities of lipogram and glycemic control finding.

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Mahmoud Abdelwahab, PhD, Study Chair — Lecturer
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ashtari S, Pourhoseingholi MA, Zali MR. Non-alcohol fatty liver disease in Asia: Prevention and planning. World J Hepatol. 2015 Jul 8;7(13):1788-96. doi: 10.4254/wjh.v7.i13.1788. PMID 26167252
- [Background] Ekstedt M, Franzen LE, Mathiesen UL, Thorelius L, Holmqvist M, Bodemar G, Kechagias S. Long-term follow-up of patients with NAFLD and elevated liver enzymes. Hepatology. 2006 Oct;44(4):865-73. doi: 10.1002/hep.21327. PMID 17006923
- [Background] Review Team; LaBrecque DR, Abbas Z, Anania F, Ferenci P, Khan AG, Goh KL, Hamid SS, Isakov V, Lizarzabal M, Penaranda MM, Ramos JF, Sarin S, Stimac D, Thomson AB, Umar M, Krabshuis J, LeMair A; World Gastroenterology Organisation. World Gastroenterology Organisation global guidelines: Nonalcoholic fatty liver disease and nonalcoholic steatohepatitis. J Clin Gastroenterol. 2014 Jul;48(6):467-73. doi: 10.1097/MCG.0000000000000116. No abstract available. PMID 24921212
- [Background] Fan JG, Kim SU, Wong VW. New trends on obesity and NAFLD in Asia. J Hepatol. 2017 Oct;67(4):862-873. doi: 10.1016/j.jhep.2017.06.003. Epub 2017 Jun 19. PMID 28642059
- [Background] Targher G, Byrne CD, Lonardo A, Zoppini G, Barbui C. Non-alcoholic fatty liver disease and risk of incident cardiovascular disease: A meta-analysis. J Hepatol. 2016 Sep;65(3):589-600. doi: 10.1016/j.jhep.2016.05.013. Epub 2016 May 17. PMID 27212244
- [Background] Younossi ZM, Gramlich T, Matteoni CA, Boparai N, McCullough AJ. Nonalcoholic fatty liver disease in patients with type 2 diabetes. Clin Gastroenterol Hepatol. 2004 Mar;2(3):262-5. doi: 10.1016/s1542-3565(04)00014-x. PMID 15017611
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. Diabetologia. 2016 Jun;59(6):1121-40. doi: 10.1007/s00125-016-3902-y. No abstract available. PMID 27053230
- [Background] Kwok R, Choi KC, Wong GL, Zhang Y, Chan HL, Luk AO, Shu SS, Chan AW, Yeung MW, Chan JC, Kong AP, Wong VW. Screening diabetic patients for non-alcoholic fatty liver disease with controlled attenuation parameter and liver stiffness measurements: a prospective cohort study. Gut. 2016 Aug;65(8):1359-68. doi: 10.1136/gutjnl-2015-309265. Epub 2015 Apr 14. PMID 25873639
- [Background] Wong VW, Vergniol J, Wong GL, Foucher J, Chan HL, Le Bail B, Choi PC, Kowo M, Chan AW, Merrouche W, Sung JJ, de Ledinghen V. Diagnosis of fibrosis and cirrhosis using liver stiffness measurement in nonalcoholic fatty liver disease. Hepatology. 2010 Feb;51(2):454-62. doi: 10.1002/hep.23312. PMID 20101745
- [Background] Karlas T, Petroff D, Garnov N, Bohm S, Tenckhoff H, Wittekind C, Wiese M, Schiefke I, Linder N, Schaudinn A, Busse H, Kahn T, Mossner J, Berg T, Troltzsch M, Keim V, Wiegand J. Non-invasive assessment of hepatic steatosis in patients with NAFLD using controlled attenuation parameter and 1H-MR spectroscopy. PLoS One. 2014 Mar 17;9(3):e91987. doi: 10.1371/journal.pone.0091987. eCollection 2014. PMID 24637477